CLINICAL TRIAL: NCT00848653
Title: The Electrode Configuration (ELECTION) CRT Study Including ELECTION Phrenic Nerve Stimulation (PNS) Sub-Study
Brief Title: ELECTION - The Electrode Configuration Cardiac Resynchronization Therapy (CRT) Study (ELECTION)
Acronym: ELECTION
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Responsible Party: Anne Swearingen, Guidant
Other Study IDs: ELECTION
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CRT device — market approved CRT device

SUMMARY:
The ELECtrode configuraTION CRT Study (ELECTION)

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is an accepted treatment for selected heart failure patients. This therapy is delivered using a device (pacemaker (PM) +/- defibrillator (ICD) ) and leads placed in the right atrium (RA), right ventricle (RV) and left ventricle (LV). Rates of LV lead implantation failure and post operative lead related have decreased dramatically over the years, however, the incidence of lead dislodgement and phrenic nerve stimulation is still high. This study is a prospective evaluation of the benefits of having various pace/sense electrode configurations available in a CRT system.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for a Guidant system, symptomatic heart failure, LV dysfunction, QRS width > 120 ms, > or = 18 yrs, able to understand the procedure, available for follow-up.

Exclusion Criteria:

* < 18 years, life expectancy < 6 months, expectation of heart transplantation during the study period, patients who have or are likely to receive a mechanical tricuspid valve, documented aortic stenosis, hypertrophic obstructive cardiomyopathy, inability or refusal to complete the follow-up at an approved centre, enrollment in another cardiovascular clinical investigation unless approved by the Manager of Clinical Studies, Guidant Canada, inability or refusal to sign consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients indicated for CRT therapy
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2004-11; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to test and compare all available LV pacing and sensing configurations | 6 months

SECONDARY OUTCOMES:
to track all programming changes made to the LV pacing/sensing configurations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Champagne, MD, Principal Investigator — Hopital Laval

REFERENCES:
- [Derived] Champagne J, Healey JS, Krahn AD, Philippon F, Gurevitz O, Swearingen A, Glikson M; ELECTION Investigators. The effect of electronic repositioning on left ventricular pacing and phrenic nerve stimulation. Europace. 2011 Mar;13(3):409-15. doi: 10.1093/europace/euq499. Epub 2011 Jan 26. PMID 21273196